CLINICAL TRIAL: NCT02738216
Title: Efficacy of a Prenatal Yoga Intervention for Antenatal Depression
Brief Title: Wellness for 2: Understanding How to Foster Well Being for Mom and Her Baby
Acronym: WF2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD081868 (NIH)
Record Dates: First submitted 2016-04-11; First posted 2016-04-14 (Estimated); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Pregnancy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prenatal Yoga (Experimental): A 9-week prenatal yoga program
  Interventions: Behavioral: Prenatal Yoga
- Mother Baby Wellness Workshop (Active Comparator): A 9-week workshop on mother and baby wellness in the first postpartum year
  Interventions: Behavioral: Mother Baby Wellness

INTERVENTIONS:
Behavioral: Prenatal Yoga — As part of the yoga program, participants will be asked to go to one 75-minute prenatal yoga class each week for 9 weeks. The yoga classes will be designed to be safe for pregnant women. In addition to classes, the yoga teacher will ask them to practice yoga at home during the program. Each participant will be given a yoga mat and a prenatal yoga DVD to take home.
  Arms: Prenatal Yoga
Behavioral: Mother Baby Wellness — This workshop is aimed at promoting moms' and babies' good health and will involve attending one 75-minute class each week for 9 weeks. Classes will cover topics such as: child development in the first year, child eating and sleeping in the first year, maintaining good health as a mom of an infant, and recent advances in women's healthcare. In addition to classes, participants will be given materials to review/ read at home.
  Arms: Mother Baby Wellness Workshop

SUMMARY:
This NICHD-funded RCT will enroll up to 178 depressed pregnant women, randomly assigning them to one of 2 intervention conditions: (1) a gentle prenatal yoga program (PYP), or (2) a series of educational workshops focused on perinatal health, the Mom and Baby Wellness Workshop (MBWW), each condition lasting 9 weeks. The investigators will clinically monitor all participants in the study for safety and clinical deterioration, and measure a variety of symptom outcomes over the course of the intervention period during pregnancy, as well as at a postpartum follow-up.

DETAILED DESCRIPTION:
In this randomized controlled trial, eligible women will be randomly assigned to either a 9-week Prenatal Yoga Program (PYP) vs. a 9-week health education control group, the Mother-Baby Wellness Workshop (MBWW). Follow up assessments will take place at multiple points during the study. The primary study outcome will be severity of prenatal depression assessed by a blind interviewer. The investigators will examine relevant secondary outcomes (self-reported depression, anxiety, functioning, & pain; pre-term birth) and potential mediators (inflammation, mindfulness/non-judgment).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy singleton pregnancy, 12-27 weeks gestation
2. Medically cleared for moderate exercise
3. Depression symptoms in moderate range. Participants must have an Quick Inventory of Depressive Symptoms (QIDS; [119]) score between 8-20
4. English-speaking
5. Aged 18 or older

Exclusion Criteria:

1. New or unstable depression treatment
2. Currently a regular yoga practitioner
3. Bipolar disorder, schizophrenia, psychotic depression, chronic psychosis
4. Current hazardous drug or alcohol use
5. Acute suicidality

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2022-11 (Actual); Study Completion 2022-11 (Actual)

PRIMARY OUTCOMES:
Quick Inventory of Depression Symptoms - Clinician Rating | Baseline to 9-week end point
  Clinician-rated depression severity

SECONDARY OUTCOMES:
Edinburgh Postnatal Depression Screen | Baseline to 9-week endpoint
  Self-reported depression severity
State-Trait Anxiety Inventory | Baseline to 9-week endpoint
  Anxiety level
Pittsburgh Sleep Quality Index | Baseline to 9-week endpoint
  Sleep disturbance
Maternal & Neonatal Outcomes Checklist (MNOC) | 30 days postpartum
  rates of preterm birth

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Battle, PhD, Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No